CLINICAL TRIAL: NCT02902783
Title: DONATE-Pilot Study: Prospective Observational Study of the ICU Management of Deceased Organ Donors
Brief Title: DONATE-Pilot Study on ICU Management of Deceased Organ Donors
Acronym: DONATE-Pilot
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Critical Care Trials Group (Other); Canadian National Transplant Research Program (Other)
Responsible Party: Sponsor
Other Study IDs: DONATE-Pilot 14-803
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-02

CONDITIONS: Deceased Organ Donors; Critical Care
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Consented deceased organ donors: Data will be collected on deceased donors, declared by neurological determination of death (DND) and by circulatory determination of death (DCD).
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Data collection relevant to this study will be obtained by observation and review of hospital charts. Limited data will be obtained through relevant organ donation organizations (ODOs).

SUMMARY:
The DONATE-Pilot is a prospective observational cohort study in organ donation (OD) that observes the ICU management of consented deceased organ donors at 4 high volume centres over a period of 12 months each. The pilot study will be followed by a 1-year prospective national observational study a 15-20 ICUs across Canada.

DETAILED DESCRIPTION:
This prospective observational cohort pilot study enrols consented organ donors admitted to 4 high volume centres over a period of 12 months. Various clinical data on deceased donors are collected prospectively from the time of consent for organ donation up to and including the day of organ recovery.

The main objectives of the DONATE-Pilot reflect the objectives of the national study which correspond to the steps in developing a platform for future clinical trials.

1. Form research teams at participating ICUs that will include an ICU physician-researcher, a local organ donation champion, ICU research coordinators and (in a limited role) a local coordinator from the provincial Organ Donation Organization (ODO);
2. Observe, record, and describe ICU practices in deceased donor care (e.g., donor resuscitation, organ suitability assessments, death declaration) which are likely to vary by site, region and province and will be very important to inform clinical care protocols for future RCTs.
3. Engage and work with ODOs from each province to foster data sharing and develop procedures to enhance efficiency in future RCTs.
4. Investigate the comparative effectiveness of various ICU interventions in deceased donor care (e.g. the potential for hormonal therapies to improve transplant rates, the potential of heparin therapy to improve peri-operative graft function);
5. Produce specific knowledge translation tools that will serve in the future as both clinical tools to enhance ICU care and research tools to facilitate future RCTs.

As part of the DONATE-Pilot we also aim to assess feasibility. Specifically the objectives are to:

1. Refine data collection procedures for deceased donors in ICU;
2. Estimate time requirements for data collection;
3. Develop efficient links to post-transplantation data and;
4. Share data as it accrues with clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a critical care area (ICU, PICU, CCU, ER)
* Consented deceased organ donors (DND and DCD)

Exclusion Criteria:

* Neonate <36 weeks gestation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients for whom consent for deceased organ donation has been obtained.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Feasibility | After 1 year of recruitment at each participating site
  This outcome is judged based on four elements: 1) Implementation of a waived consent model; 2) Refinement of data collection procedures for adult intensive care units; 3) Development of efficient links to post-transplantation data.

SECONDARY OUTCOMES:
Description of current practices | After 1 year of recruitment at each participating site
  A descriptive analysis of various interventions and approaches in the management of deceased organ donors. Adherence to recommendations of the national deceased donor management guidelines.
Effectiveness of various ICU interventions | After 1 year of recruitment at each participating site
  Defined as: 1) Number of organs recovered; 2) Number of organs transplanted.

CONTACTS AND LOCATIONS:
Overall Officials: Meade Maureen, MD, MSc, Study Director — McMaster University; Frederick D'Aragon, MD, MSc, Principal Investigator — Université de Sherbrooke
Locations (2):
- Canada (2):
  - Hamilton General Hospital, Hamilton, Ontario
  - Centre de recherche CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Aragon F, Cook D, Dhanani S, Ribic C, Burns KEA, Akhtar A, Hand L, Arseneau E, Cupido C, Whittigham H, Healey A, Frenette AJ, Lamontagne F, Meade MO; Canadian Critical Care Trials Group and the Canadian National Transplant Research Program. Hamilton-DONATE: a city-wide pilot observational study of the ICU management of deceased organ donors. Can J Anaesth. 2018 Oct;65(10):1110-1119. doi: 10.1007/s12630-018-1179-y. Epub 2018 Jul 9. PMID 29987806
- See also: DONATE Reseearch Progam Website — http://donate.ccctg.ca